CLINICAL TRIAL: NCT07302776
Title: TACTICAL: TACrolimus Targeted Immunosuppression Cessation in ALlogeneic HCT
Brief Title: TACrolimus Targeted Immunosuppression Cessation in ALlogeneic HCT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eurofins Viracor Biopharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-82367
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: GVHD; Hematopoietic Cell Transplantation (HCT); Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes; Myelofibrosis (MF); Chronic Myeloid Leukemia (CML); Chronic Myelomonocytic Leukemia (CMML)
Keywords: Post-Hematopoietic Cell Transplant (HCT) tacrolimus; hematopoietic cell transplantation (HCT)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Primary Myelofibrosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Risk-Adapted Early Tacrolimus Taper Strategy (Experimental): Initial tacrolimus dosing will be as per Standard of Care protocol. Tacrolimus is initiated at day 5 post-HCT at with initial dosing as described in Section 6.2.3, and converted to oral formulation as soon as appropriate level is achieved and the patient are able to tolerate oral dosing. Oral tacrolimus is dosed in 0.5mg increments up to two times daily. Tacrolimus levels are assessed up to three times weekly in the inpatient or outpatient setting starting 1 - 3 days after initiation to target a level of 5 - 10 ng/mL. Trough levels will be assessed as close to 12 (twice daily dosing) or 24 (daily dosing) hours as feasible after most recent dose.
  Starting on day 60, patients on Stratum A will taper tacrolimus by approximately 20% of pre-taper dose per week, rounded to the nearest 0.5 mg. Participants who meet criteria and will be completely off tacrolimus by day 88 (+/- 5 days).
  Interventions: Drug: Tacrolimus; Other: Early Tacrolimus Taper Strategy

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus is initiated on Day 5 post-HCT and transitioned to oral dosing once therapeutic levels are achieved. Oral tacrolimus is given in 0.5 mg increments up to twice daily. Levels are monitored several times weekly to target a trough of 5-10 ng/mL.
Other: Early Tacrolimus Taper Strategy — Eligible participants begin a taper on Day 60 (±5 days), reducing the tacrolimus dose by ~20% weekly, rounded to 0.5 mg, with planned discontinuation by Day 88 (±5 days). Tapering stops if significant acute GVHD develops or if unsafe.

SUMMARY:
The purpose of this study is to test the feasibility and safety of early cessation of tacrolimus following allogeneic hematopoietic cell transplantation (HCT). Post-HCT tacrolimus is given to prevent graft-vs-host-disease (GVHD), but with the use of post-transplant cyclophosphamide (PTCy), the modern approach to GVHD prevention, GVHD rates have reduced markedly.

ELIGIBILITY:
Inclusion Criteria:

* Eligible diseases:

  * Acute myeloid leukemia (AML) in complete remission (CR), CR with incomplete hematologic recovery (CRi), or MLFS.
  * Myelodysplasic syndrome (MDS) myelodysplastic syndromes eligible for alloHSCT based on IPSS-M of intermediate or higher, or IPSS-R of intermediate or higher, or refractory disease to standard growth factor or hypomethylating agent-based therapy
  * Myelofibrosis (MF)
  * Chronic myeloid leukemia (CML) in chronic phase with a prior history of accelerated phase or blast crisis or CML in chronic phase refractory to standard TKI therapy
  * Chronic myelomonocytic leukemia (CMML)
* Age ≥ 18 and ≤ 80 years at the time of enrollment.
* Planned for first myeloablative or reduced intensity allogenic transplant using a conditioning regimen listed in Appendix B.
* Has a related or unrelated donor available who is 8/8 HLA match at HLA-A, -B, -C, and -DRB1, all typed using DNA-based high-resolution methods.
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/minute or creatinine < 2 mg/dL.

Cardiac ejection fraction at rest ≥ 45% or shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA).

* Diffusing capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) ≥ 50%.
* Total bilirubin < 2 times upper limit of normal (ULN) (patients with Gilbert's syndrome may be included once hemolysis has been excluded).
* Karnofsky Performance Score ≥70%
* Negative serum or urine beta-HCG test in females of childbearing potential (FCBP) within 3 weeks of enrollment.

A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

-Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Prior allogeneic HCT.
* Planned donor lymphocyte infusion (DLI).
* Recipient positive anti-donor HLA antibodies against a mismatched allele in the selected donor determined by either:

  1. Positive crossmatch test of any titer (by complement-dependent cytotoxicity or flow cytometric testing), or
  2. Presence of anti-donor HLA antibody to any of the following HLA loci: HLA-A, -B, -C, -DRB1, -DQB1, -DQA1, -DPB1, or -DPA1, with mean fluorescence intensity (MFI) >1000 by solid phase immunoassay.
* Uncontrolled bacterial, viral, or fungal infections at time of enrollment including known, active tuberculosis infection.
* Seropositive for HIV-1 or -2, HTLV-1 or -2, Hepatitis B sAg, and/or Hepatitis C antibody.

  *History of hepatitis B or hepatitis C is permitted if viral load is undetectable per quantitative PCR and/or NAT.

Known allergy or hypersensitivity to planned GVHD prophylactic medications including PTCy, tacrolimus

* Any uncontrolled autoimmune disease requiring active immunosuppressive treatment.
* Concurrent malignancy diagnosed within 12 months of enrollment, except non-melanoma skin cancers or other early-stage solid tumors that have been curatively resected or treated to curative intent. Patients with history of low grade concurrent blood cancers that are controlled will be eligible.
* Females of childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use effective forms of birth control or abstinence for one year after transplantation.

(FCBP definition: A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

-Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the recipient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results.

* All subject files must include supporting documentation to confirm subject eligibility.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility of Early Tacrolimus Discontinuation | Day 0 through Day 180 post-transplant
  Proportion of patients who are low risk for acute graft-versus-host disease (aGVHD) who are able to discontinue tacrolimus by day 88 and who do not develop moderate to severe aGVHD by day 180.

SECONDARY OUTCOMES:
Incidence and Severity of Chronic Graft-Versus-Host Disease | Through 1 year after transplantation
  Proportion of participants who develop chronic graft-versus-host disease, reported as all grades and severe chronic graft-versus-host disease.
Incidence of Non-Relapse Mortality | 1 year post-HCT
  Incidence of death without relapse of the underlying disease.
Incidence of Disease Relapse | Through 1 year after transplantation
  Proportion of participants who experience relapse of their underlying disease.
Overall Survival | Through 1 year after transplantation
  Survival from the time of transplantation to death from any cause.
Relapse-Free Survival | Through 1 year after transplantation
  Time from transplantation to relapse of the underlying disease or death from any cause.
Graft-Versus-Host Disease-Free, Relapse-Free Survival | Through 1 year after transplantation
  Time to the first occurrence of grade III through IV acute graft-versus-host disease, chronic graft-versus-host disease requiring systemic therapy, relapse, or death.
Incidence and Severity of Infectious Complications | Through 1 year after transplantation
  Proportion of participants who develop infectious complications, reported as all grades, grade 2 through 3, and grade 3.
Incidence and Severity of Acute Graft-Versus-Host Disease | Through Day 180 after transplantation
  Proportion of participants who develop acute graft-versus-host disease, reported as all grades, grade II through IV, and grade III through IV.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States